CLINICAL TRIAL: NCT02732626
Title: The Low Voltage Guided Ablation Trial of Persistent Atrial Fibrillation
Acronym: ERASE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mödling Hospital (Other)
Collaborators: Technische Universität Dresden (Other); Medical University of Vienna (Other); Medical University of Lublin (Other); Elisabethinen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERASE V1.3
Record Dates: First submitted 2016-03-23; First posted 2016-04-08 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pulmonary vein isolation alone (Active Comparator): patients randomized to this group receive stand alone pulmonary vein isolation regardless to their left atrial voltage map
  Interventions: Procedure: radiofrequency ablation
- pulmonary vein isolation + low voltage area guided ablation (Experimental): patients randomized to this group receive pulmonary vein isolation + low voltage area guided linear substrate modification in the case if there are any
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation

SUMMARY:
This study evaluates if the exclusion of left atrial low voltage areas / scars by ablation lines in addition to pulmonary vein isolation may improve the outcome in patients with persistent atrial fibrillation in comparison to stand alone pulmonary vein isolation.

DETAILED DESCRIPTION:
This is a prospective, randomized multi center study comparing two catheter ablation strategies (pulmonary vein isolation (PVI) versus PVI plus low voltage areas (LVA) guided for ablation in patients with symptomatic persistent and long standing persistent atrial fibrillation (AF) who were unresponsive to at least one Class I or III antiarrhythmic agents, or it is the patient´s decision to receive ablation as first line therapy. Patients with documented persistent AF who are eligible for participation in the study, and gave a written informed consent, will be randomized between two groups prior to the procedure: PVI and PVI+LVAs guided radiofrequency catheter ablation.

All the patients will receive a high density voltage map in sinus rhythm (SR). All the patients will receive circumferential PVI. If LVAs are present, Patients randomized to the PVI+LVA group will get additional linear ablation lines to exclude these areas from normal voltage atrial myocardium. The patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with persistent AF documented by 12 lead ECGs (Persistent AF is defined as an AF episode which lasts longer than 7 days, Persistent AF which lasted longer than 12 months will be defined as long standing persistent AF.)
* Age 18 - 80 years, both genders
* Patient is willing to participate in the study (signed written informed consent)
* Patient is willing and available to perform all follow ups.

Exclusion Criteria:

* Atrial fibrillation due to reversible causes
* Any contraindication for AF ablation
* Contraindications to anticoagulation
* CVA/TIA in the past 6 months
* Previous left atrial catheter ablation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2016-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
recurrence of atrial arrhythmia | 12 months
  recurrence of the first symptomatic or asymptomatic episode of atrial arrhythmia within 12 months after single catheter ablation procedure, with three-month blanking

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint | 12 months
  recurrence of the first symptomatic or asymptomatic episode of atrial arrhythmia within 12 months after single catheter ablation procedure, with three-month blanking, on implanted cardiac monitors exclusively
Secondary Safety Endpoint | 90 days
  occurrence of one or more of the following adverse events within 90 days from ablation: cardiac tamponade/hemopericardium/effusion, pericarditis, stroke/TIA/arterial embolism, pulmonary vein stenosis, atrioesophageal fistula, septicemia, internal bleeding, phrenic nerve palsy, femoral vascular access complication, death

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Piorkowski, MD, Principal Investigator — Heart Center Dresden
Locations (6):
- Austria (3):
  - Moedling Hospital, Mödling, Lower Austria
  - Elisabethinen Hospital, Linz, Upper Austria
  - Landesklinikum Wiener Neustadt, Vienna
- Germany (2):
  - Heart Center Dresden, Dresden, Saxony
  - Sana Kliniken Lübeck, Lübeck
- Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huo Y, Gaspar T, Schonbauer R, Wojcik M, Fiedler L, Roithinger FX, Martinek M, Purerfellner H, Kirstein B, Richter U, Ulbrich S, Mayer J, Krahnefeld O, Agdirlioglu T, Zedda A, Piorkowski J, Piorkowski C. Low-Voltage Myocardium-Guided Ablation Trial of Persistent Atrial Fibrillation. NEJM Evid. 2022 Nov;1(11):EVIDoa2200141. doi: 10.1056/EVIDoa2200141. Epub 2022 Oct 19. PMID 38319851